CLINICAL TRIAL: NCT04373252
Title: Fecal Microbiota Transplant as a Treatment for Severe Motility Disorder
Brief Title: FMT as a Treatment for Severe Motility Disorder
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Source of FMT preps is no longer able to provide us with necessary preps.
Sponsor: University of Colorado, Denver (Other)
Collaborators: OpenBiome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-2327
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Severe Motility Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplant (Experimental): All participants will receive two fecal microbiota transplants one week apart. The transplant will occur via antegrade enema and the enema transplant material will be provided by OpenBiome, the product used is FMT Lower Delivery (FMP 30).
  Interventions: Biological: FMT Lower Delivery (FMP 30)

INTERVENTIONS:
Biological: FMT Lower Delivery (FMP 30) — Participants will receive two fecal microbiota transplants via antegrade enema, one week apart.

SUMMARY:
Many patients that are treated with anorectal malformations are fecally incontinent for life. A Bowel Management Program has been developed to help these patients by creating a daily enema regimen to keep them artificially clean of stool in the underwear. Due to the high success rate of the program, many patients who suffer from fecal incontinence due to other reasons such as, spina bifida, sacrococcygeal teratoma and sacral agenesis are referred to the program. A new issue is emerging with a group of patients that no longer obtain effective results from their daily enemas, even though they have worked successfully for years. These same patients are presenting with a narrow, spastic left colon and remarkably dilated right colon. Our hypothesis is that prolonged enema administration negatively impacts the microbiota of the colon causing the lack of response from enema administration. The purpose of this study is to restore the normal flora of the colon by fecal microbiota transplant (FMT) which we believe will improve responsiveness to enemas. By restoring colonic flora, patients will again become responsive to daily enemas and regain successful bowel management.

ELIGIBILITY:
Inclusion Criteria:

* The study population to be enrolled in this study will include patients 18 years of age and older, with a Malone (appendicostomy) or with a cecostomy, that have received daily enemas for the treatment of fecal incontinence with prior good results for months to years. However, now these patients report not having an acceptable enema response (up to 4 hours for evacuation) despite numerous attempts to adjust the enema additives. The patients typically display a narrow, spastic left colon and a dilated right colon on contrast enema. A minimum of 10 adult subjects will be enrolled first and followed for safety and efficacy outcomes for at least one month. After the initial 10 adult subjects, there will be a pause in enrollment to allow for a formal review of the adult safety and efficacy data by the primary investigator. At this time a request will be made to open enrollment of this study up to the pediatric population as well as adults.

Exclusion Criteria:

* Any patient who does not meet the above criteria will be excluded from this study. Also excluded: pregnant women, women of child-bearing potential who are unwilling to use an effective form of contraception for 30 days after FMT, women who are breastfeeding, subjects with end stage liver disease or cirrhosis, subjects with a life expectancy of less than 6 months, subjects with an absolute neutrophil count <500 cells/µL and those with severe food allergies.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Patients become responsive to daily enema treatments again | 1 year
  The primary outcome measure for this study will be the results reported in the daily journals which will identify if patients become responsive to enema treatments again (administration and complete evacuation within a one-hour period) and are able to remain clean in the underwear for 24 hours.

SECONDARY OUTCOMES:
Microbiota Analysis | 10 days
  A secondary outcome measure will come from the microbiota analysis done on the collected stool samples. By comparing the microbiota before and after FMT we will be able to determine if, and how much, the fecal microbiota transplant altered the flora of the colon.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bischoff, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No